CLINICAL TRIAL: NCT07027358
Title: Clinical Investigation Evaluating the Use of NETSmart Solution , Incorporated to NETSoins Software, in the Care and Support of Elderly People Living in Nursing Homes
Acronym: NETSMART DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Teranga Software (Industry)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A00812-45
Record Dates: First submitted 2025-05-19; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pressure Injury; Fall Prevention; Undernutrition; Drug Interaction
MeSH Terms: conditions — Pressure Ulcer; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NETSmart (Experimental): Use of NETSmart software by healthcare professionals for these patients
  Interventions: Device: NETSmart software

INTERVENTIONS:
Device: NETSmart software — Use of NETSmart software by healthcare professionals

SUMMARY:
NETSmart software is designed to help doctors, nurses and care assistants adapt the care of elderly people living in nursing homes to the following risks:

* pressure injuries
* undernutrition
* interactions between different drugs
* falls. The software analyzes the information in your medical records, alerts your medical team to any points of vigilance, and suggests appropriate recommendations.

The study comprises 2 distinct phases:

* An initial 4-month phase, during which the medical staff will simply assess whether the NETSmart software's recommendations are relevant, without changing their current practice, i.e. they will continue to care for you as usual;
* A second 6-month phase, during which your caregivers will follow the software's recommendations if they feel they are relevant, and potentially adapt your care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 70 years old
* Permanent resident at an investigation site for at least 6 months.
* Considered an at-risk patient, i.e. meeting at least one of the following criteria :
* Braden score < 16
* At risk of pressure ulcer according to the investigator's judgment
* At risk of undernutrition as judged by the investigator
* Undergoing at least 6 drug treatments
* At risk of falls as judged by the investigator
* Affiliated with the French social security system
* Having given informed, dated and signed consent to participate in the investigation

Exclusion Criteria:

* Patient with a life expectancy of less than 2 months as judged by the investigator
* Patient who is participating or has participated in another investigation or study involving the use of a medical device or drug within 30 days prior to inclusion

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of clinically relevant recommandations provided by NETSmart | 4 months
  NETSmart Software provides recommendations to the healthcare professionals. The healthcare professionals are able to mention in the software whether the recommandations are clinically relevant or not. Data will be extracted from the software to analyze this primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Maison de Famille Bourgogne, Étang-sur-Arroux, France